CLINICAL TRIAL: NCT03229590
Title: Safe Surgical Dislocation in Slipped Capital Femoral Epiphysis
Brief Title: Slipped Capital Femoral Epiphysis Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim, Principal Investigator, Assiut University
Other Study IDs: SCFE
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: SCFE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical dislocation: Reduction of slipped epiphysis via surgical dislocation technique
  Interventions: Procedure: Surgical dislocation

INTERVENTIONS:
Procedure: Surgical dislocation — Reduction of slipped epiphysis by surgical dislocation

SUMMARY:
Slipped capital femoral epiphysis represents approximately 10.8 cases per 100,000 children. The primary source for the blood supply of the head of the femur is the deep branch of the medial femoral circumflex artery. Loder described a classification for Slipped capital femoral epiphysis based on ability of the child to walk or not(walking=stable, non-walking=unstable).

DETAILED DESCRIPTION:
In slipped capital femoral epiphyses (SCFE), the severity of slippage correlates with poor long-term clinical outcome scores and radiographic evidence of osteoarthritis . In situ fixation of higher-grade SCFE has a low surgical risk and has been advocated by authors who believe the deformed hip has the potential to remodel with some restoration of the disturbed anatomic axes ; however, the remodeling potential remains controversial . Despite remodeling, the head-neck offset will remain abnormal . This is the cause of potential impingement of the femoral neck with the acetabular cartilage . Impingement in SCFE has been associated with damage of the acetabular cartilage, which may explain the early onset of osteoarthritis after SCFE .

Ganz et al. described a technique of surgical dislocation of hip involving trochanteric flip osteotomy and anterior capsulotomy preserving the blood supply to femoral head. The technique is based on extensive study of blood supply to the proximal femur. This technique allows us to completely dislocate the joint which allows complete access to intra articular pathology and allow reduction of the slipped capital femoral epiphysis .

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients with moderate Slipped capital femoral epiphysis 2- Patients with severe Slipped capital femoral epiphysis

Exclusion Criteria:

* Patients with mild Slipped capital femoral epiphysis

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The purpose of this study is to evaluate management Of moderate and severe degrees Slipped capital femoral epiphysis cases by using surgical dislocation technique .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 6 months
  this is a score for post operative evaluation of the hip (it is evaluate pain, support, Distance walked, Limp, Activities - shoes, socks, Stairs, Public transportation, Sitting, Range of motion) every item take a number then the summation of all numbers which ranged from 0 to 100 : <70 Poor 70 - 79 Fair 80-89 Good 90 -100 Excellent

REFERENCES:
- [Background] Song MH, Jang WY, Park MS, Yoo WJ, Choi IH, Cho TJ. Slipped capital femoral epiphysis in children younger than 10 years old: clinical characteristics and efficacy of physeal-sparing procedures. J Pediatr Orthop B. 2018 Sep;27(5):379-386. doi: 10.1097/BPB.0000000000000485. PMID 28704299